CLINICAL TRIAL: NCT06865794
Title: Impact of Plastic and Aesthetic Surgery on Self-esteem, a Prospective Multicentre Study
Brief Title: Impact of Plastic and Aesthetic Surgery on Self-esteem
Acronym: QUALIPLAST
Status: Not yet recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL25_0154; 2025-A00418-41 (Other: ID-RCB)
Record Dates: First submitted 2025-03-04; First posted 2025-03-10 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Self Esteem
Keywords: plastic surgery; cosmetic surgery; aesthetic surgery
MeSH Terms: interventions — Surveys and Questionnaires; Restraint, Physical

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (15):
- Breast augmentation: Adult female patient undergoing breast augmentation for aesthetic reason
  Interventions: Other: Questionnaire and Physical Exam
- Breast reduction: Adult female patient undergoing breast reduction for aesthetic reason
  Interventions: Other: Questionnaire and Physical Exam
- Mastopexy: Adult female patient undergoing Mastopexy (Breast lift) for aesthetic reason
  Interventions: Other: Questionnaire and Physical Exam
- Facelift: Adult patient undergoing facelift for aesthetic reason
  Interventions: Other: Questionnaire and Physical Exam
- Otoplasty: Adult patient undergoing otoplasty for aesthetic reason
  Interventions: Other: Questionnaire and Physical Exam
- Rhinoplasty: Adult patient undergoing rhinoplasty for aesthetic reason
  Interventions: Other: Questionnaire and Physical Exam
- Blepharoplasty: Adult patient undergoing blepharoplasty for aesthetic reason
  Interventions: Other: Questionnaire and Physical Exam
- Abdominoplasty: Adult patient undergoing abdominoplasty for aesthetic reason
  Interventions: Other: Questionnaire and Physical Exam
- Brachioplasty: Adult patient undergoing brachioplasty for aesthetic reason
  Interventions: Other: Questionnaire and Physical Exam
- Thigh lift: Adult patient undergoing thigh lift for aesthetic reason
  Interventions: Other: Questionnaire and Physical Exam
- Liposuction: Adult patient undergoing liposuction for aesthetic reason
  Interventions: Other: Questionnaire and Physical Exam
- Gender affirmation: breast augmentation: Adult patient undergoing breast augmentation gender affirmation surgery.
  Interventions: Other: Questionnaire and Physical Exam
- Gender affirmation: facial feminisation: Adult patient undergoing facial feminisation gender affirmation surgery
  Interventions: Other: Questionnaire and Physical Exam
- Gender affirmation : thoracoplasty: Adult patient undergoing thoracoplasty gender affirmation surgery
  Interventions: Other: Questionnaire and Physical Exam
- Injectables/Fillers: Adult patient undergoing Botox or Hyaluronic acid injections for aesthetic reason
  Interventions: Other: Questionnaire and Physical Exam

INTERVENTIONS:
Other: Questionnaire and Physical Exam — Rosenberg self-esteem scale pre-operatively, at 3 and 12 months post-op
  Other Names: Rosenberg self-esteem scale
Other: Questionnaire and Physical Exam — FACE-Q psychological sub-scale pre-operatively, at 3 and 12 months post-op
  Other Names: FACE-Q psychological sub-scale
  Groups: Blepharoplasty; Facelift; Injectables/Fillers; Otoplasty; Rhinoplasty
Other: Questionnaire and Physical Exam — BREAST-Q psychological sub-scale pre-operatively, at 3 and 12 months post-op
  Other Names: BREAST-Q psychological sub-scale
  Groups: Breast augmentation; Breast reduction; Mastopexy
Other: Questionnaire and Physical Exam — BSIQ-SF pre-operatively, at 3 and 12 months post-op
  Other Names: BSIQ-SF (short-form version of the Body Self-Image Questionnaire)
  Groups: Abdominoplasty; Brachioplasty; Liposuction; Thigh lift
Other: Questionnaire and Physical Exam — FLZ psychological sub-scale pre-operatively, at 3 and 12 months post-op
  Other Names: FLZ (Fragen zur Lebenszufriedenheit / Questions on Life Satisfaction) psychological sub-scale
  Groups: Gender affirmation : thoracoplasty; Gender affirmation: breast augmentation; Gender affirmation: facial feminisation

SUMMARY:
The primary objective of QUALIPLAST is to evaluate the impact of plastic and aesthetic surgery interventions on patients' self-esteem. While the demand for these procedures is steadily increasing worldwide, patients' motivations often extend beyond purely aesthetic concerns, encompassing significant psychological and emotional expectations. However, despite the growing popularity of these interventions, scientific literature remains limited when it comes to the systematic and long-term evaluation of their effects on patients' self-esteem and overall well-being.

The majority of existing studies focus on short-term outcomes or functional and physical aspects, often overlooking the psychological and emotional dimensions that play a crucial role in post-operative satisfaction. Furthermore, much research is limited to specific procedures, without adopting a comprehensive approach to plastic and aesthetic surgery. This lack of robust and generalisable data hinders a full understanding of how these interventions influence self-esteem across different types of surgeries and patient profiles.

QUALIPLAST stands out due to its multicentric, prospective, and large-scale nature, involving a wide range of procedures and collecting longitudinal data before the intervention, as well as at 3 and 12 months post-operatively. It will allow for the observation of self-esteem changes over time, providing a more complete and nuanced understanding of the effects of surgery.

This project relies on standardized and validated measurement tools, such as the Rosenberg Self-Esteem Scale, to ensure the reliability and comparability of the results. By addressing the current gaps in the literature, QUALIPLAST aims not only to enrich scientific knowledge in this field but also to provide valuable insights for healthcare professionals to improve patient care and tailor clinical practices based on the identified psychological needs.

ELIGIBILITY:
Inclusion Criteria:

Patients consulting a plastic surgeon for one of the following operations:

* Breast augmentation
* Breast reduction
* Breast lift
* Facelift
* Otoplasty
* Rhinoplasty
* Blepharoplasty
* Abdominoplasty
* Brachioplasty
* Cruroplasty
* Liposuction
* Gender affirmation: breast augmentation
* Gender affirmation: Facial feminisation
* Gender affirmation: Thoracoplasty
* Botox / Hyaluronic acid

Patients who agreed to take part in the study

Exclusion Criteria:

* Pregnant, parturient or breastfeeding women
* Minors
* Persons deprived of their liberty by a judicial or administrative decision
* Persons receiving psychiatric care
* Persons admitted to a healthcare or social institution for purposes other than research
* Adults under a legal protection measure (guardianship, curators)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Patients consulting a plastic surgeon for one of the following operations :
  * Breast augmentation
  * Breast reduction
  * Breast lift
  * Facelift
  * Otoplasty
  * Rhinoplasty
  * Blepharoplasty
  * Abdominoplasty
  * Brachioplasty
  * Cruroplasty
  * Liposuction
  * Gender affirmation: breast augmentation
  * Gender affirmation: Facial feminisation
  * Gender affirmation: Thoracoplasty
  * Botox / Hyaluronic acid
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2025-04-15 (Estimated); Primary Completion 2027-10-15 (Estimated); Study Completion 2027-10-15 (Estimated)

PRIMARY OUTCOMES:
Self-esteem score assessed by the Rosenberg self-esteem scale | Pre-operatively, at 3 and 12 months post-op
  Self-esteem score assessed by the Rosenberg self-esteem scale

CONTACTS AND LOCATIONS:
Overall Officials: Hugo Despert, Principal Investigator — Hospices Civils of Lyon
Locations (2):
- France (2):
  - Consultation Office of Dr. Emmanuel DELAY, Lyon
  - Hospices Civils of Lyon - Croix-Rousse hospital, Lyon